CLINICAL TRIAL: NCT05085184
Title: A Randomized, Open, Single-dose, 2x2x4 Replicate Crossover-design Clinical Trial to Evaluate the Safety and Pharmacokinetic Characteristics After Co-administration of UIC201806 and UIC201602 or Administration of UI018 in Healthy Volunteers
Brief Title: Study to Evaluate the Safety and PK of UI018
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korea United Pharm. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KUP-UI018-103
Record Dates: First submitted 2021-09-27; First posted 2021-10-20 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Hyperlipemia, Mixed
MeSH Terms: conditions — Hyperlipoproteinemia Type V

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- UI018 (Experimental)
  Interventions: Drug: administration of UI018
- UIC201806 and UIC201602 (Active Comparator)
  Interventions: Drug: co-administration of UIC201806 and UIC201602

INTERVENTIONS:
Drug: administration of UI018 — Test
  Arms: UI018
Drug: co-administration of UIC201806 and UIC201602 — Reference
  Arms: UIC201806 and UIC201602

SUMMARY:
This Study is to evaluate the safety and pharmacokinetics of a fixed dose combination formulation and co-administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between the ages of 19 and 45 years at screening
* Subjects whose body weight over 55 kg and ranged ± 20% of calculated Ideal body Weight(IBW) [ IBW (kg) = (height(cm) - 100) x 0.9 ]
* Subjects able to read and understand a written informed consent, and willing to decide to participate in the study.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-09-05 (Estimated)

PRIMARY OUTCOMES:
maximum concentration(Cmax) | 0 to 96 hrs
area under the curve(AUC) | 0 to 96 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Injin Jang, Dr., Principal Investigator — Seoul National University College of Medicine and Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided